CLINICAL TRIAL: NCT00002590
Title: A Pilot Study For The Treatment of Newly-Diagnosed Disseminated Anaplastic Large Cell Ki-1 Lymphoma and T-Large Cell Lymphoma
Brief Title: Combination Chemotherapy in Treating Children With Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5941; CCG-5941 (Other: Children's Cancer Group); CDR0000063751 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
Keywords: stage IV childhood lymphoblastic lymphoma; stage IV childhood large cell lymphoma
MeSH Terms: conditions — Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Cytarabine; Daunorubicin; Doxorubicin; Etoposide; Leucovorin; Methotrexate; pegaspargase; Prednisone; Thioguanine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regimen A (Experimental): See detailed description.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: thioguanine; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
  Other Names: G-CSF; Neupogen; NSC-614629
Drug: cyclophosphamide
  Other Names: Cytoxan
Drug: cytarabine
  Other Names: Cytosine Arabinoside; Ara-C; Cytosar-U; NSC-63878
Drug: daunorubicin hydrochloride
  Other Names: Daunomycin; Cerubidine
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC-123127
Drug: etoposide
  Other Names: VP-16; VePesid); NSC-141540
Drug: leucovorin calcium
  Other Names: Citrovorum Factor; Folinic Acid
Drug: methotrexate
Drug: pegaspargase
  Other Names: PEG Asparaginase; Oncaspar®
Drug: prednisone
  Other Names: NSC-10023
Drug: thioguanine
  Other Names: 6-Thioguanine; 6-TG; NSC-752
Drug: vincristine sulfate
  Other Names: Oncovin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating children who have lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the toxicity and feasibility of intensifying the New York I (NYI) regimen by adding etoposide and cytarabine, increasing the dose of methotrexate, using pegaspargase, and compressing the treatment duration (11 months) in previously untreated children with disseminated anaplastic (Ki-1 positive) large cell and large cell T-cell lymphoma. II. Provide preliminary data for a future phase III study that will compare this intensified regimen with the high-risk ALL regimen NYI in children with disseminated lymphoblastic lymphoma. III. Continue to investigate the immunophenotype, cytogenetics, and molecular biology of lymphoblastic lymphoma and their relationship to leukemia. IV. Obtain preliminary data on treatment of anaplastic large cell (Ki-1) and T-cell large cell lymphoma treated with intensive NYI.

OUTLINE: Patients with CNS disease at diagnosis receive craniospinal irradiation on Regimen A at the conclusion of Maintenance chemotherapy. The following acronyms are used: ARA-C Cytarabine, NSC-63878 CF Leucovorin calcium, NSC-3590 CTX Cyclophosphamide, NSC-26271 DNR Daunorubicin, NSC-82151 DOX Doxorubicin, NSC-123127 G-CSF Granulocyte Colony-Stimulating Factor (Amgen), NSC-614629 MTX Methotrexate, NSC-740 PEG-ASP Pegaspargase, NSC-624239 PRED Prednisone, NSC-10023 TG Thioguanine, NSC-752 VCR Vincristine, NSC-67574 VP-16 Etoposide, NSC-141540 Induction: 5-Drug Combination Systemic Chemotherapy with Hematopoietic Stimulation plus 2-Drug Combination Intrathecal Chemotherapy. VCR/PRED/CTX/DNR/PEG-ASP; with G-CSF; plus IT ARA-C/IT MTX. Consolidation: 7-Drug Combination Systemic Chemotherapy with Hematopoietic Stimulation plus Single-Agent Intrathecal Chemotherapy. VCR/PRED/PEG-ASP/VP-16/TG/ARA-C/MTX/CF; with G-CSF; plus IT MTX. Maintenance: Sequential Pulses of 2-, 3-, 3-, and 2-Drug Systemic Chemotherapy Combinations plus Single-Agent Intrathecal Chemotherapy. CTX/TG/IT MTX; VCR/PRED/DOX; VCR/MTX/CF/PEG-ASP; ARA-C/VP-16. Regimen A: Radiotherapy. Craniospinal irradiation using megavoltage equipment.

PROJECTED ACCRUAL: 40 patients will be entered over approximately 10 months. If 4 or more toxic deaths occur in the first 15 patients or 5 or more toxic deaths occur in the first 30 patients, accrual will stop. As of 05/96, asparaginase has been replaced with pegaspargase; 15-25 additional patients will be accrued. As of 01/97, a maximum of 35 patients will be accrued for PEG asparaginase-containing treatment regimen. As of 5/97, this study is open only to patients with anaplastic large cell and T cell large cell lymphoma. Approximately 60-90 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed and previously untreated anaplastic large cell Ki-1 lymphoma and T-cell large cell lymphoma Malignant lymphoblasts (identified by immunophenotype) in pleural fluid, ascitic fluid, or bone marrow sufficient for diagnosis Large cell lymphoma with T-cell phenotype eligible Localized mediastinal disease and bone lymphoma eligible CNS disease eligible and defined as: Any clearly identifiable tumor cells in cerebral spinal fluid Cranial nerve palsy (if not explained by extra cranial tumor) Clinical Spinal Cord Compression Isolated intra cerebral mass No cranial nerve palsies requiring immediate CNS irradiation

PATIENT CHARACTERISTICS: Age: Under 21 Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: Shortening fraction greater than 27% on echocardiogram (ECHO) OR Left ventricular ejection fraction greater than 47% on radionuclide scan (RCNA) OR Cardiac function assessed as within normal limits by cardiologist ECHO or RCNA obtained as close as clinically possible to start of therapy

PRIOR CONCURRENT THERAPY: No prior therapy except emergency treatment of airway obstruction or superior vena cava syndrome No more than 72 hours between emergency radiotherapy or steroids and initiation of protocol therapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 1994-07; Primary Completion 2001-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Estimate toxicity and feasibility of 11 month multiagent chemotx
  Estimate the toxicity and feasibility of a short (11 month) aggressive multiagent chemotherapy regimen - Intensive NYI\NHL

SECONDARY OUTCOMES:
Provide preliminary data for a future phase III study
Investigate the biology of lymphoblastic lymphoma
  To continue to investigate the biology of lymphoblastic lymphoma and its relationship to leukemia through the study of immunophenotyping, cytogenetics and molecular analysis.
Obtain preliminary data on treatment of anaplastic large cell
  To obtain preliminary data on treatment of anaplastic large cell (Ki-1) and T-cell large cell lymphoma treated with intensive NYI.

CONTACTS AND LOCATIONS:
Overall Officials: Minnie Abromowitch, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (33):
- United States (30):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Grace Health Centre, Halifax, Nova Scotia

REFERENCES:
- [Background] Lones MA, Perkins SL, Sposto R, Tedeschi N, Kadin ME, Kjeldsberg CR, Wilson JF, Zwick DL, Cairo MS. Non-Hodgkin's lymphoma arising in bone in children and adolescents is associated with an excellent outcome: a Children's Cancer Group report. J Clin Oncol. 2002 May 1;20(9):2293-301. doi: 10.1200/JCO.2002.06.017. PMID 11981000
- [Result] Lowe EJ, Sposto R, Perkins SL, Gross TG, Finlay J, Zwick D, Abromowitch M; Children's Cancer Group Study 5941. Intensive chemotherapy for systemic anaplastic large cell lymphoma in children and adolescents: final results of Children's Cancer Group Study 5941. Pediatr Blood Cancer. 2009 Mar;52(3):335-9. doi: 10.1002/pbc.21817. PMID 18985718
- [Result] Abromowitch M, Sposto R, Perkins S, Zwick D, Siegel S, Finlay J, Cairo MS; Children's Oncology Group. Shortened intensified multi-agent chemotherapy and non-cross resistant maintenance therapy for advanced lymphoblastic lymphoma in children and adolescents: report from the Children's Oncology Group. Br J Haematol. 2008 Oct;143(2):261-7. doi: 10.1111/j.1365-2141.2008.07320.x. Epub 2008 Aug 28. PMID 18759768
- [Result] Abromowitch M, Sposto R, Perkins S, et al.: Outcome of Children's Cancer Group (CCG) 5941: a pilot study for the treatment of newly diagnosed pediatric patients with disseminated lymphoblastic lymphoma. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A2295, 2000.